CLINICAL TRIAL: NCT00457158
Title: PREPIC 2 : Interruption of Inferior Vena Cava by a Retrievable Filter for the Prevention of Recurrent Pulmonary Embolism : a Randomised, Open Label Study
Brief Title: PREPIC 2 : Prevention of Recurrent Pulmonary Embolism by Vena Cava Interruption
Acronym: PREPIC2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government); Fondation de France (Other); Fondation de l'Avenir (Other); ALN Implants Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0501105; 2006-01-001
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Embolism; Venous Thrombosis
Keywords: pulmonary embolism; inferior vena cava filters; venous thrombosis; randomized controlled trial
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ALN optional filter
  Interventions: Device: ALN optional filter
- 2 (No Intervention): No ALN optional filter

INTERVENTIONS:
Device: ALN optional filter — J1 : ALN optional filter M3 : ALN optional filter removed
  Arms: 1

SUMMARY:
The purpose of this study is to assess efficacy and safety of optional vena cava filter implanted 3 months in prevention of recurrent pulmonary embolism in patients presenting with acute pulmonary embolism associated with thrombotic risk factors

DETAILED DESCRIPTION:
Pulmonary embolism is a common pathology, which could be fatal (about 10 000 death/year in France). It mainly originates from a deep vein thrombosis. In order to reduce mortality, prevention of new or recurrent PE is a major therapeutic aim. Only one randomised trial (PREPIC) assessed the interest of a vena cava filter in patients treated by anticoagulant treatment for a deep vein thrombosis (DVT). Results show a significant 50 % reduction of the embolic risk with the filter. This benefit occurs from the first days, but are counterbalanced by a long-term increasing risk of recurrent DVT. The filter appears promising in patients with a high risk of PE, for exemple the elderly, presenting with a thromboembolic history, cancer, heart failure or respiratory insufficiency, or a recent PE. Moreover, retrievable filters, which may be either left in place permanently or retrieved after some days or weeks, could limit the filter thrombosis risk.

The aim of PREPIC 2 study is to assess, in a multicenter randomised trial, efficacy and safety of a retrievable vena cava filter implanted 3 months versus no filter in 400 patients treated with anticoagulant drugs for a symptomatic PE associated with at least one thrombotic risk factor. A clinical follow-up will be performed at 6 months. The primary outcome is the incidence of recurrent PE at 3 months, including symptomatic and fatal PE. It will be adjudicated by an independent committee, blinded to patients' allocation.

This study will assess the benefit risk ratio of the retrievable filter for the prevention of recurrent PE, without increasing the thrombotic risk and the disadvantage due to post thrombotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Acute symptomatic pulmonary embolism; AND
* Deep or superficial vein thrombosis; AND
* At least one of the risk factors below :

  * More than 75 years old
  * Evolutiv cancer (excepting locally cutaneous cancer)
  * Known chronic heart failure treated
  * Chronic respiratory insufficiency treated
  * Bilateral deep vein thrombosis
  * Ilio-cava thrombosis
  * Ischemic stroke > 3 days and < 6 months, with lower limb deficit
  * Cardiac repercussion of pulmonary embolism assessed by echocardiography or increasing troponin I or T, or Brain Natriuretic Peptid or proBNP

Exclusion Criteria:

* Contrindication to an anticoagulant treatment or recurrent thromboembolic event despite adequate anticoagulation
* Vena cava filter already inserted
* Filter insertion impossible due to caval thrombosis
* More than 72 hours pre-randomized treatment with therapeutic dosage of anticoagulant therapy
* Non carcinologic surgery within 3 months prior randomization
* Carcinologic surgery within 10 days prior randomization
* Hypersensitivity to contrast media
* Access port in place or programmed within 3 months
* Woman who are child bearing
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2006-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
at 3 months, combined criteria including recurrent PE confirmed by objective tests and fatal PE confirmed by autopsy and death which can not be attribuated to a documented cause and for which PE/DVT can't be ruled out | 3 months

SECONDARY OUTCOMES:
recurrent pulmonary embolism, fatal or not, at 6 months (combined criteria including recurrent pulmonary ambolism confirmed by objective tests and fatal PE confirmed by autopsy and death which can not be attribuated to a documented cause and for which P | 6 months
current or new symptomatic DVT confirmed by objective tests | 6 months
mecanical complication of filter (migration, tilt, transfixion) and or puncture site hematoma, and/or local or general infection due to filter | 6 months
filter thrombosis | 6 months
filter retrieval failure | 6 months
total death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (20):
- France (20):
  - Service de Médecine Vasculaire, CHU Amiens, Amiens
  - Service d'Accueil des Urgences, CHU d'Angers, Angers
  - Service de Cardiologie, CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - Département de Medecine Interne et Pneumologie, CHU de Brest, Brest
  - Service de Pneumologie, Hôpital Antoine Beclere, Clamart
  - Service d'Accueil des Urgences, CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - Service des Urgences, CHG de Firminy, Firminy
  - Unité de Médecine Vasculaire, CHU de Grenoble, Grenoble
  - Service d'Urgences Soins Intensifs cardiologiques, CHU de Lille, Lille
  - Hôpital Edouard Herriot, Lyon
  - Service de Medecine Interne et Maladies Vasculaires, CHU de Montpellier, Montpellier
  - Service de Medecine Interne et Vasculaire, CHU de Nancy, Nancy
  - Service de Cardiologie, CHU de Nice, Nice
  - Département de Pneumologie, Hôpital Européen Georges Pompidou, AP HP, Paris
  - Service d'Urgences et de Réanimation Medicale, CHU de Saint-Etienne, Saint-Etienne
  - Service de Medecine et Therapeutique - CHU de Saint-Etienne, Saint-Etienne
  - Service de Médecine Vasculaire, CH Toulon, Toulon
  - Service de Cardiologie, CHU de Tours, Tours

REFERENCES:
- [Background] Decousus H, Leizorovicz A, Parent F, Page Y, Tardy B, Girard P, Laporte S, Faivre R, Charbonnier B, Barral FG, Huet Y, Simonneau G. A clinical trial of vena caval filters in the prevention of pulmonary embolism in patients with proximal deep-vein thrombosis. Prevention du Risque d'Embolie Pulmonaire par Interruption Cave Study Group. N Engl J Med. 1998 Feb 12;338(7):409-15. doi: 10.1056/NEJM199802123380701. PMID 9459643
- [Background] PREPIC Study Group. Eight-year follow-up of patients with permanent vena cava filters in the prevention of pulmonary embolism: the PREPIC (Prevention du Risque d'Embolie Pulmonaire par Interruption Cave) randomized study. Circulation. 2005 Jul 19;112(3):416-22. doi: 10.1161/CIRCULATIONAHA.104.512834. Epub 2005 Jul 11. PMID 16009794
- [Derived] Mismetti P, Laporte S, Pellerin O, Ennezat PV, Couturaud F, Elias A, Falvo N, Meneveau N, Quere I, Roy PM, Sanchez O, Schmidt J, Seinturier C, Sevestre MA, Beregi JP, Tardy B, Lacroix P, Presles E, Leizorovicz A, Decousus H, Barral FG, Meyer G; PREPIC2 Study Group. Effect of a retrievable inferior vena cava filter plus anticoagulation vs anticoagulation alone on risk of recurrent pulmonary embolism: a randomized clinical trial. JAMA. 2015 Apr 28;313(16):1627-35. doi: 10.1001/jama.2015.3780. PMID 25919526